CLINICAL TRIAL: NCT06798922
Title: Flap Sparing in Postoperative Radiotherapy of Oral Cavity Cancers: a De-escalation Randomized Phase III Trial
Brief Title: Flap Sparing in Postoperative Radiotherapy of Oral Cavity Cancers
Acronym: OPTIFLAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A01764-43
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Oral Cavity Carcinoma; Flap; Radiotherapy, Adjuvant; Reconstruction Surgery
Keywords: protontherapy; flap; oral cavity carnicoma; radiotherapy; IMRT
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (Active Comparator): Standard IMRT or proton therapy practice, usual CTV definition
  Interventions: Radiation: Standard post-operative radiotherapy without flap sparing (current practice)
- Experimental arm (Experimental): IMRT or proton therapy with flap sparing
  Interventions: Radiation: Post-operative radiotherapy with flap sparing

INTERVENTIONS:
Radiation: Standard post-operative radiotherapy without flap sparing (current practice) — Standard post-operative radiotherapy without flap sparing (current practice)
  Arms: Standard arm
Radiation: Post-operative radiotherapy with flap sparing — Post-operative radiotherapy with flap sparing
  Arms: Experimental arm

SUMMARY:
Patients with oral cavity cancer treated by reconstructive surgery with a flap.

Patients will be treated in the study for :

* Experimental arm: Post-operative radiotherapy with flap sparing
* Control arm: Standard post-operative radiotherapy without flap sparing (current practice) Radiotherapy by IMRT using photons or proton therapy (IMPT)

DETAILED DESCRIPTION:
Patients with oral cavity cancer treated by reconstructive surgery with a flap.

Patients will be treated in the study for :

* Experimental arm: Post-operative radiotherapy with flap sparing
* Control arm: Standard post-operative radiotherapy without flap sparing (current practice) Radiotherapy by IMRT using photons or proton therapy (IMPT) Our purpose is to demonstrate the feasibility of sparing surgical flaps from radiotherapy, in order to reduce toxicity while maintaining local disease control.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Performance Status 0-2
* Patient with oral cavity cancer (soft tissue or soft tissue-bone flap), treated by reconstructive surgery with a flap. Oropharynx cancer whose flap extends significantly into the oral cavity may be included in the study
* Quality of resection with margins > 1 mm
* Patient candidate to post-operative radiotherapy (Intensity-Modulated Radiation Therapy (IMRT) or proton therapy)
* Concomitant chemotherapy is allowed (stratification parameter)
* Patient must have signed a written informed consent form prior to any trial specific procedures
* Patient affiliated to the social security system

Exclusion Criteria:

* Local flap (small size limiting IMRT modulation potential)
* History of radiotherapy of head and neck area
* Metastatic disease
* History of other malignancy within the previous 3 years (except for appropriately treated in-situ cervix carcinoma and non-melanoma skin carcinoma)
* Simultaneous participation in another clinical study may compromise the conduct of this study.
* Pregnant or lactating women
* Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
* Patient deprived of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2034-03-01 (Estimated)

PRIMARY OUTCOMES:
loco-regional control rate | 2 years after the end of postoperative radiotherapy
  To evaluate whether flap sparing yields non-inferior 2-year loco-regional control rate as flap-agnostic radiotherapy (as per standard routine practice) in completely resected oral cavity carcinomas undergoing postoperative radiotherapy

SECONDARY OUTCOMES:
Proportion of patients with acute and late Ear-Nose-Throat (ENT) toxicities | within 12 months after postoperative radiotherapy
  Rate of Ear-Nose-Throat (ENT) toxicities among cavity cancer patients with a flap, defined as the proportion of oral cavity cancer patients with at least two ENT toxicities grade ≥ 2 according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (24):
- France (24):
  - Chu Amiens, Amiens
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre François Baclesse, Caen
  - CHU CAEN, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHIC, Créteil
  - Centre Georges-François Leclerc, Dijon
  - Centre Guillaume le Conquérant, Le Havre
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - APHM Marseille, Marseille
  - Institut Régional du Cancer Val D'aurelle, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - Centre Antoine Lacassagne, Nice
  - APHP La Pitié, Paris
  - Chu Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Chu Rouen, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - IUCT, Toulouse
  - Chu Tours, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Thariat J, Leconte A, Lequesne J, Vela A, Carsuzaa F, Dejean C, Renard S, Pereira S, Lebars S, Nadin L, Plisson L, Bastit V, Woisard V, Hervieu-Klisnick Z, Lasne-Cardon A, Clarisse B. Flap sparing in postoperative radiotherapy versus standard flap-agnostic radiotherapy of oral cavity cancers (OPTIFLAP): protocol for a de-escalation, randomised, non-inferiority, phase III trial. BMJ Open. 2025 Sep 14;15(9):e109094. doi: 10.1136/bmjopen-2025-109094. PMID 40953868